CLINICAL TRIAL: NCT05792254
Title: Efficacy and Safety of Huaier Granule in Patients With Stage I Primary Ovarian Fallopian Tube Cancer After Peritoneal Cancer: a Single-center Prospective Single-arm Study
Brief Title: Huaier Granule in Patients With Stage I Primary Ovarian Fallopian Tube Cancer After Peritoneal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023(01)
Record Dates: First submitted 2023-01-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-01

CONDITIONS: Primary Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Huaier granule (Experimental): Huaier granule is supplied as 20-g granule. Huaier granule will be administered as 20 g orally tid x 28 days (continuous). One cycle = 28 days. There is no planned treatment interruption between cycles. In the absence of intolerable toxicity, a patient may continue to receive treatment with Huaier granule until disease progression, or until 24 months have elapsed.
  Interventions: Drug: Huaier granule

INTERVENTIONS:
Drug: Huaier granule — Oral Huai Er granules, 20 g once, 3 times a day, continued to progress or intolerance toxicity.

SUMMARY:
This study is an exploratory, single-center, prospective single-arm study to explore the efficacy of Huaier granules in the treatment of stage Ⅱ-Ⅳ primary ovarian cancer, fallopian tube cancer, and peritoneal cancer after satisfactory tumor reduction (R0/R1). Twenty-five patients with FIGOⅡ-Ⅳ ovarian cancer, peritoneal cancer or tubal cancer confirmed by histopathology were enrolled and treated with Huaier granules. During the study period, the patients were followed up once at 3 months, and the medication was continued until progression or intolerability of toxicity. This is an exploratory, single-center, prospective single-arm study to explore the efficacy of Huaier granules in the treatment of stage Ⅱ-Ⅳ primary ovarian cancer, fallopian tube cancer, and peritoneal cancer after satisfactory tumor reduction (R0/R1). Twenty-five patients with FIGOⅡ-Ⅳ ovarian cancer, peritoneal cancer or tubal cancer confirmed by histopathology were enrolled and treated with Huaier granules. During the study period, the patients were followed up once at 3 months, and the medication was continued until progression or intolerability of toxicity.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of Huai er granule in the treatment of stage I primary ovarian cancer, fallopian tube cancer and peritoneal cancer

Secondary objectives:

1. To analyze the safety of Huaier granule in the treatment of ovarian fallopian tube cancer and peritoneal cancer after operation;
2. To analyze the influence of Huaier granule on the quality of life of postoperative patients with ovarian fallopian tube cancer and peritoneal cancer

Exploratory objective:

To evaluate the efficacy of Huaier granule in patients with BRCA mutation and BRCA wild-type ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

1. ≥18years old
2. Histopathologically confirmed FIGO II-IV stage primary ovarian cancer peritoneal or fallopian tube cancer
3. Patients who underwent primary tumor reduction or intermediate tumor reduction with satisfactory results (R0/R1) within 15 days after surgery
4. After tumor reduction, the physician assessed that chemotherapy was not suitable or the patient was unwilling to receive chemotherapy
5. Life expectancy is 3 months
6. Liver and kidney function :

   1. AST and ALT 3 times the upper limit of normal value or 5 times the upper limit of normal value in the presence of liver metastasis; T
   2. he upper limit of total bilirubin 3 times normal value;
   3. Serum creatinine is 3 times the upper limit of normal
7. No other tumors, no history of other malignant tumors (except non-melanoma skin cancer in situ cervical cancer or other cancers that have received curative treatment and have no signs of disease for at least 5 years)
8. Voluntarily participate in the study and sign the informed consent

Exclusion Criteria:

1. Breastfeeding women during pregnancy
2. Recurrent ovarian cancer
3. Known allergy to the study drug;
4. Central nervous system diseases or brain metastases;
5. History of abdominal/pelvic radiotherapy;
6. History of organ transplantation history of immune deficiency disease requiring systemic steroid therapy or other immunosuppressive therapy
7. Hiv-ag /AB test result is positive;
8. Complicated with serious cardiovascular and cerebrovascular diseases or other serious diseases affecting follow-up treatment of subjects: such as myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months; Uncontrolled hypertension after antihypertensive therapy (systolic ≥140 or diastolic ≥90 mmHg); Uncontrolled diabetes mellitus (HbA1c>8.0%) etc
9. Participate in other clinical study patients within 1 month
10. Poor compliance is estimated to be difficult to complete the follow-up
11. In addition to the above, the investigator determined that the patients were not suitable for the clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival rate | up to 1 years from start of treatment
  The time from study entry to the time of disease progression as determined by the investigator (by clinical, radiological or pathological means) or death from any cause

SECONDARY OUTCOMES:
Progression Free survival | Every 3 month until 2 years from start of treatment
  PFS according to the RECIST 1.1 criteria, based on the investigator's assessment.
1 year overall survival rate | one year
  Observed length of life from entry into the study to death; or for living patients, the date of last contact regardless of whether or not this contact is on a subsequent protocol.
Quality of life score（FACT-O） | Every 3 month until 2 years from start of treatment
  The FACT-O questionnaire consists of a Physical Well-Being Section, Social/Family Well-Being Section, Emotional Well-Being Section, Functional Well-Being Section, and Additional Concerns Section
pain score | Every 3 month until 2 years from start of treatment
  In the Visual Analog Score to be used as the pain measurement criterion, '0' indicates no pain, while '10' defines the most severe pain.
the Rates of AE and SAE | Every 3 month until 2 years from start of treatment
  frequency of adverse events according to MedDRA terms